CLINICAL TRIAL: NCT00961103
Title: Assessment of Motor Development Related to Use of Orthoses in SMA II and III
Brief Title: Motor Development and Orthoses in Spinal Muscular Atrophy (SMA)
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: UDGEE-SMA
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Spinal Muscular Atrophy
Keywords: spinal muscular atrophy; motor development; orthoses
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- SMA II and SMA III: patients with SMA II and SMA III

SUMMARY:
Spinal Muscular Atrophy (SMA) is neurodegenerative disease of anterior horn cells of spinal cord and represents the second more frequent pathology in childhood.

According to the age of onset and the maximum motor function the disorder is classified in 4 types. Patients with SMA II and SMA III often use orthoses to achieve postural and dynamic functions.

In this retrospective observational study the investigators describe the characteristics of sitting position, standing and walking correlated to type and time of orthoses used.

DETAILED DESCRIPTION:
We collect data from patients with SMA II and SMA III referred to UDGEE from jan. 1995 to dec. 2008.

We estimate to achieve informations about 50-70 patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and genetics diagnosis of SMA II and SMA III

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with SMA II and SMA III referred to UDGEE for rehabilitation consultation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-10-12 (Actual); Primary Completion 2009-11-01 (Actual); Study Completion 2011-04-04 (Actual)

PRIMARY OUTCOMES:
time and percentage of sitting, standing, walking achievement in SMA II and SMA III | aug.2009- nov.2009

SECONDARY OUTCOMES:
characteristics and percentage of orthoses for postural sitting control , standing and walking in SMA II and SMA III | aug. 2009 - dec.2009

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Ferrari, MD, Study Director — Hospital S.Maria Nuova Reggio Emilia Italy
Locations (1):
- UDGEE Hospital S.Maria Nuova, Reggio Emilia, RE, Italy

REFERENCES:
- [Background] Wang CH, Finkel RS, Bertini ES, Schroth M, Simonds A, Wong B, Aloysius A, Morrison L, Main M, Crawford TO, Trela A; Participants of the International Conference on SMA Standard of Care. Consensus statement for standard of care in spinal muscular atrophy. J Child Neurol. 2007 Aug;22(8):1027-49. doi: 10.1177/0883073807305788. PMID 17761659